CLINICAL TRIAL: NCT03491761
Title: Does Intra-articular Platelet-Rich Plasma Injection Provide Superior Outcomes Compared With Viscosupplementation in the Treatment of Knee Osteoarthritis?
Brief Title: Intra-articular Platelet-Rich Plasma Compared With Viscosupplementation in the Treatment of Knee Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Jason Koh, Board of Directors Endowed Chair of Orthopaedic Surgery, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH17-199
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: Platelet Rich Plasma (PRP); Viscosupplementation; Knee Osteoarthritis; Hyaluronic Acid (HA); WOMAC; KOOS; Euflexxa
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PRP Treatment (Experimental): PRP is injected using 22 gauge needles through the classic approach (lateral midpatellar) in a sterile setting. The PRP is obtained from a maximum 16 cc sample of the patients' blood drawn at the time of treatment. Using sterile technique, the venous blood is transferred to a centrifuge and prepared by the centrifugation process for 5 minutes. 4-7 mL of PRP is transferred from the large outer syringe into the small inner syringe and injected within 30 minutes of being spun to negate the need of anticoagulants. The procedure will take approximately 20-30 minutes.
  Interventions: Biological: PRP Treatment
- HA Treatment (Active Comparator): HA is injected using 22 gauge needles through the classic approach (lateral midpatellar) in a sterile setting. Euflexxa will be prepared according to the package insert.
  Interventions: Biological: HA Treatment

INTERVENTIONS:
Biological: PRP Treatment — PRP will be prepared using an Arthrex ACP® kit (a low-leukocyte Autologous Conditioned Plasma system). This is a single-spin system that concentrates platelets and separates red blood cells (RBCs) as well as white blood cells (WBCs) from the treatment product.
  Other Names: Platelet-Rich Plasma
  Arms: PRP Treatment
Biological: HA Treatment — Euflexxa will be used for treatment. It will be prepared according to the package insert.
  Other Names: Hyaluronic Acid; Euflexxa
  Arms: HA Treatment

SUMMARY:
This is a single-center, prospective, randomized, single-blind, comparator therapy, parallel group study for symptomatic patients diagnosed with knee osteoarthritis. The aim is to demonstrate superior efficacy of platelet-rich plasma (PRP) as compared to hyaluronic acid (HA) in treating knee osteoarthritis. This aim will be objectively measured by endpoint consisting of changes in cartilage thickness from baseline in the MRI. The Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire will be used to calculate The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score. It will measure changes in pain and function from baseline. Approximately 100 subjects will be treated at NorthShore University HealthSystem (NorthShore) as part of this study. This study has the potential to improve outcomes in a very common chronic degenerative disease, osteoarthritis, which can have a significant effect on individuals' quality of life.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, comparative clinical trial with an allocation ratio of 1:1. The primary endpoint is the MRI-based cartilage thickness measurement. The secondary endpoint is the The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score. There are 2 arms: PRP treatment and HA treatment. Due to the treatment procedure, the study will not be blinded to either the subject or PI. However, the radiologist that scores the cartilage thickness will be blinded with regard to clinical characteristics and treatment of subjects.

The subjects are randomized with 1:1 block randomization with a block size of 4 patients. The patient population is symptomatic patients diagnosed with knee osteoarthritis K-L grade 2 or 3. The sample size is 100 total subjects (50 in each arm). The duration is approximately 13 months, final data accumulated at month 12 after treatment at single site - NorthShore.

All potential subjects will complete screening blood work which will consist of a complete blood count to include platelets and differential (CBC with Diff), c-reactive protein (CRP), and a sed rate (ESR).

Patients randomized into the PRP group will also have at the time of the procedure whole blood and PRP analyzed for PLT, WBC, and RBC per injection, and a CBC with leukocyte differential will be performed on the PRP to evaluate the fold increase in platelet concentrations. The amount of blood taken for the procedure will be approximately 15 ml (3-4 teaspoons). Four to six milliliters are injected back into the knee as plasma rich platelets.

Patients randomized to the HA group will not undergo any laboratory testing.

Data will be summarized as mean±sd for continuous variables and frequencies and percentages for categorical variables. For the primary analysis, repeated measures ANOVA will be performed on both primary and secondary endpoints using baseline and 12 months data to examine the differences in changes between PRP and HA groups. In addition, linear mixed models will be used to analyze WOMAC scores (baseline, 1m, 3m, 6m, and 12m) and MRI data (baseline, 6m, 12m) using all available data collected from all time points. All analysis will be performed with SAS 9.3 (SAS Inc., Cary, NC). A p value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Chronic pain (>3 months)
* Grade 2 -3 according to Kellgren- Lawrence (K-L) classification system (using bilateral anteroposterior radiograph image acquired while the patient is weight-bearing with both knees in full extension)
* Minimum score of 40 out of possible 100 on the VAS (Visual Analog Scale) for pain
* Age 18 to 75 years old
* Physical exam and medical history
* Complete Blood Count to include platelets and differential (CBC with Diff) within normal limits
* C-Reactive Protein (CRP) within normal limits
* Sed Rate (ESR) within normal limits
* Survey of current medications

Exclusion Criteria:

* Presence of major axial deformity (>5° valgus or varus deviation)
* Surgery on target knee within 12 months prior to scheduled treatment
* Autoimmune disorder
* Active infections
* Immuno-suppression (e.g., AIDS, etc.)
* Anti-coagulant therapy
* Use of NSAIDs 5 days prior to blood draw or up to 7 days after last PRP / HA treatment
* Hemoglobin (Hg) <12 g/dL
* Platelet counts (PLT) <150,000 /mm3
* Previous infiltrative treatment within 3 weeks prior to scheduled treatment
* Pregnancy/Breastfeeding
* Hypersensitivity to HA
* Inability to complete an MRI due to metal implants or claustrophobia
* Diabetes
* Active treatment for a malignancy
* Active wound in the knee
* Recent history of knee trauma
* Vasovagal history
* An injection of hyaluronic acid (HA) or platelet-rich plasma (PRP) to the affected knee within the last two years.
* In the judgment of the investigator, the patient is unable to perform and/or complete all of the study visits or treatments required.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cartilage Thickness on MRI | 6 and 12 months
  Evaluation of changes from baseline in central medial femorotibial compartment cartilage thickness measurements (via ordered value method) using quantitative T1 and cartilage compositional changes using T2 MRI at 6 and 12 months.

SECONDARY OUTCOMES:
3. A secondary outcome will be measuring changes in the KOOS Jr (Knee injury and Osteoarthritis Outcome Score) | 6 weeks, 12 weeks, 6 months, and 12 months
  The KOOS is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score will be calculated using KOOS Questionnaire. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). The total WOMAC score is created by summing the items for all three subscales, with higher scores reflecting worse pain, stiffness, and physical function. Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
  This objective will be measured in WOMAC total score from baseline to 6 weeks, 12 weeks, 6 months, and 12 months in 100 subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Koh, MD, MBA, Principal Investigator — Clinical Chairman, Dept. of Orthopaedics
Locations (1):
- NorthShore University HealthSystems, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided